CLINICAL TRIAL: NCT02751879
Title: Real-world Data on Gi(l)Otrif® Dose Adjustment in First-line Treatment, TKI-naïve, Advanced Non-small Cell Lung Cancer Patients With EGFR Activating Mutations
Brief Title: Real World Data on Gi(l)Otrif® Dose Adjustment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.270
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Non small cell lung cancer (NSCLC): patients with Epidermal growth factor receptor (EGFR) mutation (common mutations), TKI-naïve advanced non small cell lung cancer (NSCLC), treated with Gi(l)otrif® as the first-line treatment for NSCLC within the approved label

SUMMARY:
This is a non-interventional, multi-country, multi-site study based on existing data from medical records of patients treated with Gi(l)otrif® as part of the routine treatment according to the approved label. Data from real-world will help to understand if dose modifications are done similar as in LUX-Lung 3 trial and if the outcome on safety and effectiveness are as in trial settings. Furthermore, data on modified starting doses, the underlying reasons and effects on safety and outcome are needed.

ELIGIBILITY:
Inclusion criteria:

1. Age = 18 years
2. Patients with Epidermal growth factor receptor (EGFR) mutation (common mutations), tyrosine kinase inhibitors (TKI)-naïve advanced non small cell lung cancer (NSCLC), treated with Gi(l)otrif® as the first-line treatment for NSCLC within the approved label
3. Signed and dated written informed consent per regulations. (Exemption of a written informed consent for retrospective observational studies in some countries per local regulations and legal requirements.)

Exclusion criteria:

1. Any contraindication to Gi(l)otrif® as specified in label.
2. Patients with uncommon mutations are excluded as uncommon mutations are not within label in all participating countries (e.g. USA).
3. Patients still on treatment with Gi(l)otrif® will be excluded unless treatment period is > or = 6 months.
4. Patients treated with Gi(l)otrif® within an interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (29):
- United States (2):
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
- SMZ Baumgartner Hoehe Otto Wagner Spital, Vienna, Austria
- BC Cancer Agency - Vancouver, Vancouver, British Columbia, Canada
- France (4):
  - HOP Jean Minjoz, Besançon
  - HOP Dijon, Cardio-Pneumo, Dijon, Dijon
  - HOP Européen G. Pompidou, Paris
  - HOP Tenon, Paris
- Germany (3):
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Klinikum Nürnberg, Nuremberg
  - Pius-Hospital, Oldenburg, Oldenburg
- Italy (2):
  - Azienda Ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Vito Fazzi, Lecce
- Japan (2):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Kurashiki Central Hospital, Okayama, Kurashiki
- Mexico (3):
  - Centro Medico ABC, Mexico City
  - Organización para Cuidado Integral en Oncología S.A de C.V, Monterrey
  - Unidad de Cancerologia, Zapopan
- Poland (3):
  - Medical Practice,Bogdan Zurawski,Private Practice,Bydgoszcz, Bydgoszcz
  - Grzegorz Czyzewicz Specialised Medical Practice, Cracow, Krakow
  - Greater PL Cent.Pulmo.&Thor.Surg.Eugenia&Janusz Zeyland, Poznan
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (3):
  - Yeungnam University Medical Center, Daegu
  - Chonbuk National University Hospital, Jeonju
  - Pusan National Univ. Hosp, Pusan
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona (Barcelona)
  - Hospital La Princesa, Madrid
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Halmos B, Tan EH, Soo RA, Cadranel J, Lee MK, Foucher P, Hsia TC, Hochmair M, Griesinger F, Hida T, Kim E, Melosky B, Marten A, Carcereny E. Impact of afatinib dose modification on safety and effectiveness in patients with EGFR mutation-positive advanced NSCLC: Results from a global real-world study (RealGiDo). Lung Cancer. 2019 Jan;127:103-111. doi: 10.1016/j.lungcan.2018.10.028. Epub 2018 Nov 2. PMID 30642537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a non-interventional, multi-country, multi-site study based on existing data from medical records of patients treated with Gi(l)otrif® tablet once daily as indicated in the approved labels. Between December 2016 and October 2017, 231 patients were screened for study participation and 228 patients were treated.
Pre-assignment Details: All patients were screened for eligibility to participate in the study. Patients attended specialist sites which would then ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to study if any of the specific entry criteria were violated.
Groups:
- Gi(l)Otrif ≥ 40 mg: Patients were orally treated with starting dose of greater than or equal to 40 mg Gi(l)otrif tablet once daily.
- Gi(l)Otrif ≤ 30 mg: Patients were orally treated with starting dose of less than or equal to 30 mg Gi(l)otrif tablet once daily.
Period: Overall Study
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg
Started | 157 | 71
On Treatment at Study Completion | 81 | 41
Completed | 157 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All registered patients with informed consent (as applicable with local regulations) and at least one administration of Gi(l)otrif®.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg | Total
Number analyzed (Participants) | 157 | 71 | 228
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of all patients included in the trial Population: FAS
  Years | 64.50 (12.00) | 68.10 (10.84) | 65.62 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender distribution of all patients included in the trial. Population: FAS
  Participants
    Female | 90 | 48 | 138
    Male | 67 | 23 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity of all patients included in the trial. Population: FAS
  Participants
    Hispanic or Latino | 16 | 9 | 25
    Not Hispanic or Latino | 120 | 56 | 176
    Unknown or Not Reported | 21 | 6 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of all patients included in the trial. Population: FAS
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 74 | 26 | 100
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 1 | 0 | 1
    White | 59 | 37 | 96
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 22 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Adverse Drug Reactions (ADR) by Severity Class.
Description: An adverse drug reaction (ADR) is defined as a response to a medicinal product which is noxious and unintended. Grade 1, Grade 2, Grade 3 and Grade 4 ADR severity classes were considered for assessment of this outcome.
Time Frame: From signing the informed consent onwards until the end of the study, up to 104 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients (%)
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg
Number analyzed (Participants) | 157 | 71
Percentage of patients (%)
  Grade 1 | 21.02 | 21.13
  Grade 2 | 44.59 | 57.75
  Grade 3 | 24.84 | 16.90
  Grade 4 | 3.18 | 0.00

2. Primary Outcome: Time on Treatment With Gi(l)Otrif®
Description: Time on treatment with Gi(l)otrif® in real-world setting has been calculated in this assessment. Time on treatment refers to time to treatment failure with Gi(l)otrif®
Time Frame: From first dose of Gi(l)otrif® treatment to last dose of Gi(l)otrif® treatment, up to 104 weeks.
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg
Number analyzed (Participants) | 157 | 71
Months | 18.22 [14.61 to 21.51] | 19.41 [12.93 to NA] — The upper limit of the Confidence Interval has not being reached.

3. Primary Outcome: Time to Progression With Gi(l)Otrif®
Description: Time to progression was calculated from the date of first dose of Gi(l)otrif® treatment to the earliest date of documented progression (clinical, radiographic or both clinical/radiographic progression) or tumour-related death, whatever occurred first.
Time Frame: From first dose of Gi(l)otrif® treatment to last dose of Gi(l)otrif® treatment, up to 104 weeks.
Population: FAS
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg
Number analyzed (Participants) | 157 | 71
Months | 20.03 [18.22 to 23.98] | 25.92 [17.3 to NA] — The upper limit of the Confidence Interval has not being reached.

4. Secondary Outcome: Percentage of Patients With a Modified Starting Dose of Gi(l)Otrif®
Description: Percentage of patients with a modified starting dose that is dose other than the recommended 40 mg daily of Gi(l)otrif® has been calculated to assess this outcome measure.
Time Frame: From first dose of Gi(l)otrif® treatment to last dose of Gi(l)otrif® treatment, up to 104 weeks.
Population: FAS
Measure: Number; unit: Percentage of patients (%)
Groups:
- Modified Starting Dose of Gi(l)Otrif: All patients who were treated with starting dose other than recommended dose of 40 mg Gi(l)otrif treatment once daily.
Arm/Group | Modified Starting Dose of Gi(l)Otrif
Number analyzed (Participants) | 73
Percentage of patients (%)
  50 mg | 2.74
  30 mg | 94.52
  20 mg | 2.74

5. Secondary Outcome: Percentage of Patients With Reasons for Modified Starting Dose of Gi(l)Otrif®
Description: Different reasons for starting dose with modified dose that is dose other than recommended 40 mg once daily.
Time Frame: From first dose of Gi(l)otrif® treatment to last dose of Gi(l)otrif® treatment, up to 104 weeks.
Population: FAS
Measure: Number; unit: Percentage of patients (%)
Groups:
- Modified Dose of 50 mg Gi(l)Otrif: All patients who were treated with modified dose of 50 mg Gi(l)otrif treatment once daily.
- Modified Dose of ≤ 30 mg Gi(l)Otrif: All patients who were treated with modified starting dose of less than of equal to 30 mg Gi(l)otrif treatment once daily.
Arm/Group | Modified Dose of 50 mg Gi(l)Otrif | Modified Dose of ≤ 30 mg Gi(l)Otrif
Number analyzed (Participants) | 2 | 71
Percentage of patients (%)
  Patient's condition | 0.00 | 38.03
  Previous experience with EGFR-TKI | 0.00 | 5.63
  Institutional standard | 100.00 | 15.49
  Other | 0.00 | 40.85

ADVERSE EVENTS:
Time Frame: From signing the informed consent onwards until the end of the study, up to 104 weeks.
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Full Analysis set (FAS): All registered patients with informed consent (as applicable with local regulations) and at least one administration of Gi(l) otrif® was used for this assessment. This was a single-arm retrospective analysis.
Arm/Group | Gi(l)Otrif ≥ 40 mg | Gi(l)Otrif ≤ 30 mg
All-Cause Mortality (participants affected / at risk) | 8/157 | 0/71
Serious Adverse Events (participants affected / at risk) | 11/157 | 7/71
Other Adverse Events (participants affected / at risk) | 147/157 | 68/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gi(l)Otrif ≥ 40 mg (N=157) | Gi(l)Otrif ≤ 30 mg (N=71)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gi(l)Otrif ≥ 40 mg (N=157) | Gi(l)Otrif ≤ 30 mg (N=71)
Diarrhoea (Gastrointestinal disorders) | 120 | 51
Stomatitis (Gastrointestinal disorders) | 59 | 20
Paronychia (Infections and infestations) | 79 | 39
Rash pustular (Infections and infestations) | 11 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 73 | 32
Dry skin (Skin and subcutaneous tissue disorders) | 17 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 8
Nausea (Gastrointestinal disorders) | 3 | 5
Dysgeusia (Nervous system disorders) | 2 | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
Due to non-interventional character there were no predefined examinations, retro- and prospective data could be collected, bias regarding AE documentation, participation of patients on treatment was limited due to one exclusion criterion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT02751879/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT02751879/SAP_001.pdf